CLINICAL TRIAL: NCT06534736
Title: Effects of Scapular Stabilization Exercises Combined With Post Facilitation Stretch in Patients With Upper Cross Syndrome: A Randomized Control Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/19
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Upper Cross Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups.Sample will be divided into two groups , Group A and Group B.Group A i.e Control group will receive Post Faciliation Stretch only for 4 weeks on alternative days.Group B i.e intervention hgroup will undergo Scapular Stabilization exercises along with post facilitation stretch for 4 weeks on alternative days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post Facilitation Stretch Group (Experimental): Treatment protocol given to both groups will be carried out for 3 sessions per week for 4 weeks.
  It will comprise of hot pack for 10 minutes, Tens for 10 minutes. Participants will be instructed to maintain the contraction for 6 to 10 seconds and then relax the muscles as quickly as possible.The stretch will be held for 15 seconds in an attempt to lengthen the shortened facscial structures.The muscles which will be targeted are Levator Scapular Upper Trapezius Sternocleidomastoid scalene Pectoralis Muscles
  Interventions: Procedure: Electrotherapy and physical agents; Procedure: Post Facilitation Stretch
- Stabilization Exercises along with the PFS Group (Experimental): It will comprise of hot pack for 10 minutes, Tens for 10 minutes. Participants will be instructed to maintain the contraction for 6 to 10 seconds and then relax the muscles as quickly as possible.The stretch will be held for 15 seconds in an attempt to lengthen the shortened facscial structures.The muscles which will be targeted are Levator Scapular Upper Trapezius Sternocleidomastoid scalene Pectoralis Muscles Scapular Stabilization exercises protocol will be carried out in 4 weeks , 3 sessions per week. Scapular wall slide exercise will be carried out with body weight .Scapular retraction with body weight. Wall Ball Circle exercise with body weight for the first two weeks and then with dumbbells for the next two weeks. Scapular Squeeze again with the body weight and dumbbells. Wall press ups will be performed. Post Facilitation stretch of the targeted muscles also will be carried out during the sessions
  Interventions: Procedure: Electrotherapy and physical agents; Procedure: Post Facilitation Stretch; Procedure: Scapular Stabilization Exercise

INTERVENTIONS:
Procedure: Electrotherapy and physical agents — It will comprise of hot pack for 10 minutes, Tens for 10 minutes.
Procedure: Post Facilitation Stretch — Participants will be instructed to maintain the contraction for 6 to 10 seconds and then relax the muscles as quickly as possible.The stretch will be held for 15 seconds in an attempt to lengthen the shortened facscial structures.The muscles which will be targeted are Levator Scapular Upper Trapezius Sternocleidomastoid scalene Pectoralis Muscles
Procedure: Scapular Stabilization Exercise — Scapular Stabilization exercises protocol will consist of scapular wall slide exercise, scapular retraction, wall Ball Circle exercises, scapula squeeze, wall press ups. Exercise program 3 sets of 5 - 10 repetition for 10 seconds hold a 20 second break between each sets. The intervention will be applied 2 weeks 3 times a week and 30 min per session. Post Facilitation stretch of the targeted muscles also will be carried out during the sessions
  Arms: Stabilization Exercises along with the PFS Group

SUMMARY:
Upper Cross Syndrome is characterized by the postural deviation of head , neck , shoulders and altered muscular muscular activation which included weakness of rhomboids , middle and lower trapezius and serratus anterior and tightness of upper trapezius , pectorallis and levator scapulae . It is a combinaton of scapular dyskinesia , forward head posture , rounded shoulder and thoracic kyphosis.This study aims to assess the enduring effects scapular stabilization exercises along with post facilitation stretch on Upper Cross Syndrome with the goal of preventing its reoccurrence over time, If there are improved results by the combination of both treatments than any of them alone , then it can used in combination for better results on patients

ELIGIBILITY:
Inclusion Criteria

* Aged 18 to 45 with neck pain for more than 3 months
* Both genders males and females
* NPRS scoring of greater than or equal to 4 points
* No History of serious pathology or recent neck trauma
* Diagnosed Upper Cross Syndrome cases using Janda approach

Exclusion Criteria

* Known Scapular or shoulder pathology
* Cervical and thoracic fractures , dislocations or surgeries or whiplash injury

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-12-10 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | 4 weeks
  Measured with Numeric Pain Rating Scale
Neck Disability | 4 weeks
  Neck disability index is used for assessing self-rated disability in neck pain patients
Cervical Range of Motion | 4 weeks
  Goniometer will be used to measure Cervical Range of Motion

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan